CLINICAL TRIAL: NCT07326111
Title: A Clinical Trial of Tirzepatide (LY3298176) in Subjects With Overweight or Obesity and PCOS-related Ovarian Dysfunction
Brief Title: A Clincial Study Testing Tirzepatide on Reproductive Function and Metabolic Health in Women With PCOS Who Are Overweight or Obese
Acronym: PERIODS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Bonn (Other)
Collaborators: Heart and Diabetes Center North Rhine-Westphalia (Other); University Hospital, Essen (Other); Ruhr University of Bochum (Other); LMU Klinikum (Other)
Responsible Party: Principal Investigator, Charlotte Fries, Senior Physician, University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MED1-202202; 2024-515982-32-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-09; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Polycystic Ovary Syndrome (PCOS); Obesity & Overweight
Keywords: pcos; tirzepatide; obesity; reproductive health; polycystic ovary syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity; Overweight | interventions — Tirzepatide

STUDY DESIGN:
Intervention Model Description: Multi-centre, prospective, randomized, double-blind and placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Active Comparator): Weekly abdominal subcutaneous injection of tirzepatide over a 72-week treatment period including a 20-week dose-escalating regiment and 52-week treatment period adjunct to reduced-calorie diet and increased physical activity
  Interventions: Drug: Tirzepatide as an adjunct to lifestyle intervention
- Control Group (Placebo Comparator): Weekly abdominal subcutaneous injection of a placebo injectable over a 72-week period ad-junct to reduced-calorie diet and increased physical activity.
  Interventions: Drug: Placebo as an adjunct to lifestyle intervention

INTERVENTIONS:
Drug: Tirzepatide as an adjunct to lifestyle intervention — Doses: 2.5 mg, 5 mg, 7.5 mg, 10 mg, 12.5 mg, 15 mg Mode of application: weekly subcutaneous injection, prefilled pen injector Duration of treatment: 72 weeks (20 weeks dose escalation, 52 weeks treatment with maximum tolerated dose)
  Arms: Treatment Group
Drug: Placebo as an adjunct to lifestyle intervention — Dose: Placebo Pens to mimic doses 2.5 mg, 5 mg, 7.5 mg, 10 mg, 12.5 mg, 15 mg Mode of Application: weekly subcutaneous injection, prefilled pen injector Duration of Treatment: 72 weeks
  Arms: Control Group

SUMMARY:
This clinical study examines whether tirzepatide can improve ovarian dysfunction in premenopausal women with polycystic ovary syndrome (PCOS) who are overweight or have obesity. Tirzepatide is already approved for the treatment of diabetes and obesity, but its effects on ovarian dysfunction in PCOS are not yet known. Participants will be randomly assigned to tirzepatide or placebo in a double-blinded manner.

The goal of the study is to demonstrate that tirzepatide, at the maximum tolerated dose, is superior to placebo for improvement of ovarian dysfunction as defined by menstrual irregularity in overweight or obesity-related PCOS.

All participants will have a screening visit, followed by 72 weeks of treatment. Treatment includes a 20-week dose-escalation period and a 52-week maintenance period. Lower doses may be used if side effects occur, and the highest tolerated dose will be continued through the maintenance phase. A 4-week safety follow-up will take place after treatment, and long-term follow-up will continue for one year. The study will take place at five clinical trial sites in Germany.

DETAILED DESCRIPTION:
PERIODS is a prospective, phase IV, multi-centre, randomized, double-blind and placebo-controlled clinical trial that will investigate the effects of tirzepatide compared with placebo on ovarian dysfunction in premeno-pausal, overweight (BMI ≥ 27 kg/m2) women with PCOS. The primary endpoint is the improvement of ovarian dysfunction as defined by menstrual irregularity and ovulation frequency in overweight or obesity-related PCOS.

All subjects will undergo a screening visit and a 72-week treatment period including a 20-week dose escalation up to the maximum tolerated dose. Lower doses of tirzepatide are permitted if intolerable side effects occur. However, even if a lower dose of tirzepatide turns out to be the maximum tolerated dose, this lower dose will be administered for the entire 20-week dose escalation period, followed by the 52-week maintenance dose.

The safety follow-up period will be 4 weeks (for subjects completing or discontinuing IMP during the first 72 weeks). Long-term follow-up will be one year after discontinuation of IMP.

The trial design is multi-centred with a planned number of 5 participating trial sites in Germany.

ELIGIBILITY:
General Inclusion Criteria

* Written informed consent to participate in this clinical trial in accordance with local regulations and the ethical review board governing this clinical trial
* Subjects

  * motivated, capable, and willing to self-inject IMP, as required for this protocol.
  * motivated, capable, and willing to follow trial procedures for the duration of the clinical trial, includ-ing, but not limited to lifestyle, dietary and exercise advice.
  * motivated, capable, and willing to complete trial diaries and required questionnaires.

Indication-specific Inclusion Criteria

* Females aged 18 - 45 years of childbearing potential
* At least 3 years post-menarche and premenopausal
* BMI ≥ 27 kg/m²
* Previous diagnosis of PCOS, defined by Rotterdam criteria
* Oligomenorrhea or secondary amenorrhea with irregular periods (defined as cycle length less than 21 or more than 35 days or < 8 cycles per year); within the last 10 years (if currently receiving hormonal contraceptive treatment) OR over the last year in the absence of hormonal contraceptive treatment
* Biochemical signs of hyperandrogenism with total testosterone in upper 95th Percentile AND free androgen index (FAI) > ULN and/or clinical signs of hyperandrogenism
* Hormonal contraceptive naïve or not on hormonal contraceptives six months prior to screening, willing to be without hormonal contraceptives for the duration of the clinical trial and to perform safe alternate contraception (barrier methods) during the 72-week IMP intake period and 30 days after the last dose of IMP

General Exclusion Criteria

* Subjects without legal capacity who are unable to understand the nature, scope, significance and consequences of this clinical trial
* Subjects with a physical or psychiatric condition which at the investigator's discretion may put the subject at risk, may confound the trial results, or may interfere with the subject's participation in this clinical trial

  * Note: Patients with depression or other psychiatric disorder whose disease state is considered stable and expected to remain stable throughout the course of the clinical trial, in the opinion of the investigator, may be considered for inclusion.
  * Note: Subjects with a lifetime suicidal event cannot be considered for inclusion
* Simultaneous participation in another clinical trial, or participation in a clinical trial taking an investiga-tional product, up to 30 days after last IMP intake in that clinical trial
* Known or persistent abuse of medication, drugs or alcohol
* History of an active or untreated malignancy or being in remission from a clinically significant malig-nancy for less than 5 years

  o Excluding basal- or squamous-cell skin cancer or in situ carcinomas of the cervix
* Prior diagnosis of severe renal impairment or measured as estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m² during screening
* Acute or chronic hepatitis, signs and symptoms of any other liver disease other than non-alcoholic fatty liver disease, or alanine aminotransferase (ALT) level > 3.0 X the upper limit of normal, as deter-mined by the laboratory during screening
* History of gastric emptying abnormality (e.g., gastroparesis, gastric outlet obstruction or chronic de-pendence on drugs that significantly affect gastric emptying)
* Current (positive pregnancy test, e.g., ß-HCG test in urine / serum) or planned pregnancy during the 72-week treatment period from randomization, or nursing women

Indication-specific Exclusion Criteria

* Prior diagnosis of diabetes mellitus other forms than type 2

  o Note: Excluding prior history of gestational diabetes
* In case of diabetes mellitus type 2, exclusion of subjects

  * on DPP-4 inhibitors, GLP-1R agonist and/or a dual/triple incretin agonist (up to 6 months prior to screening)
  * on sulfonylureas or insulin (basal and/or bolus)
  * with uncontrolled diabetes (HbA1c > 8.5%)
  * with non-proliferative diabetic retinopathy requiring acute treatment
  * with diabetic maculopathy
  * Note: use of metformin or SGLT-2-inhibitor (if needed for glycemic control in type-2-diabetes) is allowed
* Current or prior treatment (up to 6 months prior to screening) with GLP-1R agonist or a dual incretin agonist for obesity or other indications
* Use of inositol formulations (up to 6 months prior to screening)
* Congenital adrenal hyperplasia (CAH, classic and non-classic forms)
* Thyroid, pituitary, and/or adrenal disease (if not appropriately treated)

  o Note: Excluding stable disease and/or stable drug dose 12 weeks before screening
* Hyperprolactinaemia
* Known history of benign intrauterine lesions
* Hysterectomy
* Known history of hypersensitivity against tirzepatide or excipients
* Known history of hypersensitivity against medroxyprogesterone acetate or dydrogesterone or any other ingredients of the Auxiliary Medicinal Products
* Known personal or family history of medullary thyroid cancer or subjects with Multiple Endocrine Ne-oplasia syndrome type 2 (MEN 2)
* Elevated calcitonin levels as determined by the laboratory during screening

  * ≥ 20 ng/L, if eGFR ≥ 60 mL/min/1.73 m2
  * ≥ 35 ng/L, if eGFR < 60 mL/min/1.73 m2
* Known secondary cause of obesity (i.e., Cushing syndrome) or monogenetic or syndromic forms of obesity (i.e., melanocortin 4 receptor deficiency or Prader Willi Syndrome)
* Known history of acute or chronic pancreatitis
* Previous or planned bariatric surgery or endoscopic and/or device-based therapy for obesity

  o Note: excluding liposuction or abdominoplasty if performed > 1 year prior to screening
* Vaginal bleeding of unknown cause
* Known thromboembolic events or active thrombophlebitis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — transgender men under gender-affirming hormone therapy (GAHT) are not eligible
Enrollment: 198 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of ovarian dysfunction as defined by menstrual irregularity in overweight or obesity-related PCOS | At 72 weeks after randomization
  1. Mean menstrual bleeding ratio (number of menstrual bleedings divided by treatment period in months) during the last 52 weeks of treatment, assessed at 72 weeks after randomization
  2. Mean change in menstrual bleeding ratio from baseline, calculated at 72 weeks after randomization (with baseline defined as mean menstrual bleeding ratio during the 6 months before randomization)
Key Secondary - Improvement of ovarian dysfunction as defined by ovulation frequency in overweight or obesity-related PCOS | Within 24 weeks after completed dose titration
  Total number of biochemically confirmed ovulatory events (within 24 weeks after completed dose titration) measured by weekly serum progesterone

SECONDARY OUTCOMES:
Percentage of Participants With Normalization of Menstrual Cycle | Week 72
  Normalization of the menstrual cycle is defined as a cycle length greater than 21 days and less than 35 days, or more than 8 cycles per year. This endpoint compares the proportion of subjects achieving this criteria in the tirzepatide group versus the placebo group.
Change From Baseline in Serum Anti-Müllerian Hormone (AMH) | Baseline and Week 72
  Assessment of AMH as a surrogate marker for ovarian follicle pool and ovarian morphology.
Change From Baseline in Biochemical Androgen Profile | Baseline and Week 72
  Evaluation of the androgenic status including Total Testosterone, Sex Hormone-Binding Globulin (SHBG), DHEA-S, and Androstenedione. Results will be reported as the change from baseline or the ratio of Week 72 to baseline.
Change From Baseline in Calculated Free Androgen Index (FAI) and Calculated Free Testosterone | Baseline and Week 72
  FAI is calculated as (Total Testosterone/SHBG) x 100. Free Testosterone is calculated using the Vermeulen formula or a similar validated method based on Total Testosterone and SHBG levels.
Change From Baseline in Pituitary-Gonadal Hormones (LH, FSH, Estradiol, Progesterone) | Baseline and Week 72
  Assessment of the hormonal regulation of the ovarian cycle by measuring Luteinizing Hormone (LH), Follicle-Stimulating Hormone (FSH), Estradiol, and Progesterone.
Percentage Change in Body Weight from Baseline to Week 72 | Baseline and Week 72
  Relative change in total body weight compared to the starting weight.
Percentage of Participants Achieving ≥ 5%, ≥ 10%, ≥ 15%, and ≥ 20% Body Weight Loss | Baseline and Week 72
  Proportion of subjects in each treatment arm who reach the specified weight loss thresholds at Week 72.
Change from Baseline in Body Composition (BIA) at Week 72 | Baseline and Week 72
  Mean change in fat mass and fat-free mass as measured by Bioelectrical Impedance Analysis (BIA).
Change from Baseline in Waist Circumference and Waist-to-Hip Ratio | Baseline and Week 72
  Measurement of abdominal fat distribution change from randomization to Week 72.
Change from Baseline in Fasting Glucose and HbA1c at Week 72 | Baseline and Week 72
  Assessment of long-term and fasting glycemic control.
Change from Baseline in Systemic Insulin Sensitivity Indices | Baseline and Week 72
  Evaluation of insulin sensitivity using the Quantitative Insulin Sensitivity Check Index (QUICKI), Homeostasis Model Assessment (HOMA-IR), and Matsuda's Insulin-Sensitivity Index derived from OGTT data.
Change from Baseline in Fasting Lipid Profile at Week 72 | Baseline and Week 72
  Mean change in Triglycerides and the Triglyceride-to-HDL Ratio.
Change from Baseline in Fasting Lipid Profile at Week 72 | Baseline and Week 72
  Mean change in Total Cholesterol, LDL Cholesterol and HDL cholesterol
Change from Baseline in Liver Enzymes and Non-invasive Biomarkers (FLI, FIB-4) | Baseline and Week 72
  Assessment of liver health via Fatty Liver Index (FLI) and FIB-4 Score.
Change from Baseline in Liver Stiffness and Fat Content at Week 72 | Baseline and Week 72
  Measurement of hepatic steatosis and fibrosis via imaging (e.g., Transient Elastography/FibroScan).
Change from Baseline in Systolic and Diastolic Blood Pressure | Baseline and Week 72
  Mean change in SBP and DBP from randomization to Week 72.
Change from Baseline in High-Sensitivity C-Reactive Protein (hs-CRP) | Baseline and Week 72
  Marker for systemic meta-inflammation.
Change From Baseline in the 36-Item Short Form Survey (SF-36) at Week 72 | Baseline and Week 72
  The SF-36 is a multi-purpose, short-form health survey with 36 questions. It yields an 8-scale profile of functional health and well-being scores. Each scale is transformed to a 0-100 range, where 0 indicates the lowest level of health and 100 indicates the highest level of health (higher scores mean a better outcome).
Change From Baseline in the Polycystic Ovary Syndrome Health-Related Quality of Life Questionnaire (PCOSQ) | Baseline and Week 72
  The PCOSQ measures health-related quality of life in women with PCOS across five domains (Emotions, Body Hair, Weight, Infertility, and Menstrual Problems). Each item is scored on a 7-point scale. Domain scores range from 1 to 7, where higher scores indicate better health-related quality of life/less distress.
Change From Baseline in the European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) | Baseline and Week 72
  The EQ-5D-5L consists of a descriptive system (5 dimensions) and a Visual Analogue Scale (VAS). The VAS records the respondent's self-rated health on a vertical scale where the endpoints are labeled 'The best health you can imagine' (100) and 'The worst health you can imagine' (0). Higher scores mean a better outcome.
Patient Global Impression of Severity (PGI-S) at Week 72 | Baseline and Week 72
  The PGI-S is a single-item question asking the patient to rate the severity of their condition. It uses a 5-point scale: 1 (None), 2 (Mild), 3 (Moderate), 4 (Severe), 5 (Very Severe). A decrease in score indicates an improvement in condition.

OTHER OUTCOMES:
Dose-Dependent Menstrual Bleeding Ratio at Week 72 | Week 72
  Evaluation of the dose-response relationship of tirzepatide (5 mg, 10 mg, and 15 mg) compared to placebo. Mean menstrual bleeding ratio at 72 weeks after randomization.
Dose-Dependent Change in Mean Menstrual Bleeding Ratio at Week 72 | Baseline and Week 72
  Evaluation of the dose-response relationship of tirzepatide (5 mg, 10 mg, and 15 mg) compared to placebo. Mean change in menstrual bleeding ratio at 72 weeks after randomization
Dose-Dependent Normalization of Menstrual Cycle | 72 weeks
  Evaluation of the dose-response relationship (5 mg, 10 mg, and 15 mg) compared to placebo. Percentage of subjects achieving a cycle length > 21 and < 35 days or > 8 cycles/year.
Total Number of Biochemically Confirmed Ovulatory Events (Dose-Response) | 24 weeks following completed dose titration
  Evaluation of the dose-response relationship (5 mg, 10 mg, and 15 mg) compared to placebo. Number of ovulatory events (serum progesterone ≥ 3 ng/mL) during the 24 weeks following completed dose titration.
Change From Baseline in Ovarian Volume (MTD vs. Placebo) | 72 weeks
  Change in ovarian volume (OV) measured by transvaginal ultrasound, comparing the maximum tolerated dose (MTD) of tirzepatide to placebo.
Change From Baseline in Follicle Number Per Ovary (MTD vs. Placebo) | 72 weeks
  Change in follicle number per ovary (FNPO) measured by transvaginal ultrasound (MTD vs. placebo).
Change From Baseline in Hirsutism (Ferriman-Gallwey Score) at MTD | 72 weeks
  Assessment of hair growth using the modified Ferriman-Gallwey score. Scale: 0 (no hair) to 36 (severe hirsutism). A decrease in score indicates improvement.
Change From Baseline in Female Pattern Baldness (Ludwig Scale) at MTD | 72 weeks
  Assessment using the Ludwig scale (Grade I, II, or III). Higher grades indicate more severe hair loss. A decrease in grade indicates improvement.
Change From Baseline in Acne Lesion Count at MTD | 72 weeks
  Count of acne spots per side of the face (MTD vs. placebo).
Percentage of Participants Reaching HbA1c Targets (< 7% and < 6.5%) at MTD | 72 weeks
  Proportion of diabetic participants reaching glycemic targets (MTD vs. placebo).
Change From Baseline in HbA1c at MTD | 72 weeks
  Mean change in HbA1c (%) from randomization to Week 72 (MTD vs. placebo).
Menstrual Bleeding Ratio Within 52 Weeks After Drug Discontinuation | Week 124
  Mean bleeding ratio calculated during the off-drug period (Week 72 to Week 124).
Change in Menstrual Bleeding Ratio (Treatment vs. Follow-up) | Week 72 to Week 124
  Comparison of the bleeding ratio during the treatment phase (up to Week 72) versus the bleeding ratio during the 52-week follow-up phase (Week 124).
Percentage of Participants Maintaining Menstrual Cycle Normalization at Week 124 | Week 124
  Proportion of participants who still meet the criteria for normal cycles (21-35 days or >8/year) 52 weeks after stopping tirzepatide.
Change From Baseline in Ovarian Volume (OV) and Follicle Number (FNPO) at Week 124 | Baseline and Week 124
  Assessment of sustained effects on ovarian morphology via transvaginal ultrasound 52 weeks after drug discontinuation.
Change From Baseline in Serum Anti-Müllerian Hormone (AMH) at Week 124 | Baseline and Week 124
  Evaluation of AMH levels as a marker of ovarian reserve and morphology after the 52-week follow-up period.
Change From Baseline in Androgen Profile and Gonadotropins at Week 124 | Baseline and Week 124
  Includes Total Testosterone, Estradiol, Progesterone, SHBG, DHEA-S, Androstenedione, LH, and FSH measured 52 weeks after drug discontinuation.
Change From Baseline in Calculated Free Androgen Index (FAI) and Free Testosterone at Week 124 | Baseline and Week 124
  Calculation of FAI [(Total Testosterone/SHBG) x 100] and free testosterone to assess sustained biochemical improvement after drug discontinuation.
Sustained Improvement in Hirsutism (Ferriman-Gallwey Score) at Week 124 | Baseline and Week 124
  mFG score (range 0-36, higher score = more severe) measured 52 weeks after drug discontinuation. A lower score compared to baseline indicates sustained improvement.
Sustained Improvement in Female Pattern Baldness (Ludwig Scale) and Acne at Week 124 | Baseline and Week 124
  Assessment of hair loss (Ludwig Grade I-III) and acne lesion counts (number of spots) at the end of the follow-up period.
Clinical Pregnancy Rate at Week 124 | From Week 72 to Week 124
  Percentage of subjects who achieve clinical pregnancy (confirmed by ultrasound visualization of fetal cardiac activity) after drug discontinuation. This includes conception via natural/spontaneous means, pharmacologically induced ovulation (e.g., letrozole, clomiphene), or Assisted Reproductive Technology (ART).
Change From Baseline in Body Weight and Composition at Week 124 | Baseline and Week 124
  Mean and percentage change in body weight, fat mass, and fat-free mass (measured by BIA) 52 weeks after drug discontinuation.
Percentage of Participants Maintaining Weight Loss Thresholds at Week 124 | Week 124
  Proportion of participants maintaining ≥ 5%, ≥ 10%, ≥ 15%, and ≥ 20% weight loss from randomization at the end of the follow-up period.
Change From Baseline in Waist Circumference and Waist-to-Hip Ratio at Week 124 | Baseline and Week 124
  Assessment of abdominal fat distribution 52 weeks after drug discontinuation.
Change From Baseline in Fasting Glucose and HbA1c at Week 124 | Baseline and Week 124
  Change From Baseline in Fasting Glucose and HbA1c at Week 124
Change From Baseline in Insulin Sensitivity Indices (QUICKI, HOMA-IR, Matsuda) at Week 124 | Baseline and Week 124
  Derived from fasting and OGTT data to assess sustained effects on insulin sensitivity.
Change From Baseline in Fasting Lipid Parameters at Week 124 | Baseline and Week 124
  Assessment of sustained effects on total cholesterol, HDL and LDL cholesterol 52 weeks after drug discontinuation.
Change From Baseline in Fasting Lipid Parameters at Week 124 | Baseline and Week 124
  Assessment of sustained effects and Change From Baseline in fasting triglycerides and Triglyceride-to-HDL Cholesterol Ratio 52 weeks after drug discontinuation.
Change From Baseline in Liver Enzymes at Week 124 | Baseline and Week 124
  Mean change in serum levels of liver enzymes (e.g., ALT, AST, GGT) to assess sustained hepatic safety and function 52 weeks after drug discontinuation.
Change From Baseline in Non-invasive Liver Scores (FLI and FIB-4) at Week 124 | Baseline and Week 124
  Evaluation of the Fatty Liver Index (FLI) and the Fibrosis-4 (FIB-4) score 52 weeks after drug discontinuation.
Change From Baseline in Blood Pressure | Baseline and 124 weeks
  Assessment of sustained effects on systolic/diastolic BP
Change From Baseline in hs-CRP at Week 124 | Baseline and week 124
  Assessment of sustained effects on systemic meta-inflammation (hs-CRP).
Change From Baseline in the 36-Item Short Form Survey (SF-36) at Week 124 | Baseline and Week 124
  The SF-36 is a health survey yielding scores from 0 to 100. Higher scores indicate a better health-related quality of life. Assessment of sustained well-being 52 weeks after drug discontinuation.
Change From Baseline in the PCOS Health-Related Quality of Life Questionnaire (PCOSQ) at Week 124 | Baseline and Week 124
  The PCOSQ measures five domains (Emotions, Body Hair, Weight, Infertility, Menstrual Problems) on a scale of 1 to 7. Higher scores indicate better health-related quality of life.
Change From Baseline in EQ-5D-5L Health State Index Score at Week 124 | Baseline and Week 124
  The EQ-5D-5L Index Score is derived from 5 dimensions (Mobility, Self-care, Usual activities, Pain/discomfort, and Anxiety/depression). Each dimension has 5 levels. The scores are converted into a single index value using a country-specific value set (e.g., German Value Set). The index score ranges from less than 0 (where 0 is death) to 1 (perfect health). Higher scores indicate a better health state.
Patient Global Impression of Severity (PGI-S) at Week 124 | Week 124
  A single-item scale where patients rate their disease severity from 1 (None) to 5 (Very Severe). A decrease in score indicates improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Wiebke K. Fenske, Professor, Principal Investigator — BG UniversitätsklinikumBergmannsheil Bochum
Locations (2):
- Germany (2):
  - University Hospital BG Bergmannsheil Bochum General internal medicine, endocrinology and diabetology, gastroenterology and hepatology, Bochum
  - University Hospital Bonn Division of Endocrinology, Diabetes and Metabolism, Bonn

IPD SHARING:
Plan to Share IPD: Yes
Individual subject data will be available. Individual subject data (including data dictionaries) that underlie results concerning primary or secondary endpoints reported in a published scientific article will be shared on demand after deidentification. Furthermore, the following documents will be made available at least: Trial Protocol and Informed Consent Form. The data will be shared immediately following publication and ending 10 years following publication. Data are made available to researchers after a methodologically sound scientific proposal has been submitted to the Coordinating Investigator, and a steering committee consisting of the Coordinating Investigator, the representative of the Coordinating Investigator, and an authorized SZB member has approved the proposal. The data will be shared to achieve aims in the approved proposal.
  Proposals should be directed to Wiebke.Fenske@rub.de. To gain access, data requestors will need to sign a data access agreement.
Time Frame: The data will be shared immediately following publication and ending 10 years following publication.
Access Criteria: To gain access, data requestors will need to sign a data access agreement.